CLINICAL TRIAL: NCT03429283
Title: Achromobacter Xylosoxidans Infections : Epidemiology and Environmental Investigations
Brief Title: Achromobacter Xylosoxidans (ACHX) Infections
Acronym: ACHX
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 16/E/19
Record Dates: First submitted 2017-12-07; First posted 2018-02-12 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2018-02

CONDITIONS: Nosocomial Infection
Keywords: Epidemiology,; Achromobacter xylosoxidans,; antibiotic resistance
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive retrospective epidemiological study — descriptive retrospective epidemiological study

SUMMARY:
Data extraction from bacteriological laboratory of Martinique University hospital to determine the frequency and the distribution of nosocomial infections due to Achromobacter xylosoxidans (ACHX), an emerging multi-resistant environmental bacteria. The specific tropical environment and climatic conditions in Martinique may favor ACHX development and the investigators suppose that this new opportunistic pathogen can represent a danger for hospitalized patients. The aim of our study is to describe the most affected population and try to identify the main environmental sources of contamination.

DETAILED DESCRIPTION:
In June 2016, a patient who developed a Staphylococcus aureus mediastinitis died of a superinfection by Achromobacter xylosoxidans. This germ is an hydrotelluric bacteria described as emergent and multi-resistant, involved in nosocomial infections. It is known to be responsible for severe nosocomial infections in immunocompromised individuals (endocarditis, bacteriemia, wound infections, pneumonia) associated with high morbidity and mortality but it is also able to infect immunocompetent patients. According to literature, it is capable of developing in antiseptic and disinfectant solutions due to the acquisition of resistance to these products. Moreover it has a great ability to form biofilms, resulting in major eradication difficulties, both on the environmental and clinical level.

Various environmental sources of contamination have been identified, including dental units water lines, dialysis water, nebulizers, reusable boxes of disinfectant wipes, siphons of patient's rooms, vials of heparin...

There is no evidence for the existence of a possible portage in humans, but ACHX has already been isolated from the intestine of a 3-month-old baby who has never received antibiotic treatment. On the other hand, this germ colonizes the respiratory system of patients with cystic fibrosis. The frequency of isolation in sputum of these patients is increasing for a decade for still unknown reasons. ACHX surgical site infections are rare and to our knowledge only two cases of ACHX mediastinitis have been reported in the literature to date, either because cases are indeed rare or because the high mortality rate restricts publications. The clinical case of our CHU caught our attention and the investigators contacted the laboratory of bacteriology to inquire about the existence of other cases of infection with this germ. The investigators have then seen that ACHX seems to evolve in low noise for more than 10 years in our hospital with about 10 cases of infection per year.

Also, the investigators wanted to learn more and propose a study articulated around two axes:

* An epidemiological axis, in which the investigators detail local epidemiology, calculate rates of impact and analyze their evolution over 10 years, identify the most affected units, identify the types of most common infections, identify a population at risk, study profiles of resistance of the isolated strains,
* An environmental axis with identification of potential sources after development of appropriate analytical methods.

The ultimate goal of this study is the protection of patients by the fight against ACHX nosocomial infections and other related germs, by preventive eradication methods of environmental sources once they have been identified. The investigators want to avoid a new fatal infection episode.

A research of ACHX natural reservoirs in Martinique is also conceivable subsequently, the hypothesis being that this germ, particularly greedy of heat and humidity, is very present in a tropical environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in Martinique University Hospital, Pierre Zobda Quitman site, from January 2006 to December 2016, with biological sample positive to ACHX

Exclusion Criteria:

* Patient hospitalized in another site…
* Patients hospitalized less than 48h before bacteriological analysis……

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The incidence rate of Achromobacter xylosoxidans nosocomial infections | january 2006 to december 2016
  number of infections/ total number of patients hospitalized in our institution

SECONDARY OUTCOMES:
The incidence density of Achromobacter xylosoxidans nosocomial infections | january 2006 to december 2016
  number of infections/ total number of days of hospitalization
Mortality rate related to ACHX, | january 2006 to december 2016
  number of deaths at three months

CONTACTS AND LOCATIONS:
Overall Officials: Karine SANCHEZ, Pharma D, Principal Investigator — Martinique University Hospital
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No